CLINICAL TRIAL: NCT00573248
Title: Nicotine and Behavioral Regulation in Adult ADHD
Brief Title: Nicotine and Behavior in Adult ADHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 2005-4296; TRDRP grant# 14RT-0147H
Record Dates: First submitted 2007-12-12; First posted 2007-12-14 (Estimated); Results first posted 2011-09-02 (Estimated); Last update posted 2011-09-09 (Estimated); Status verified 2011-09

CONDITIONS: ADHD
Keywords: Nicotine; ADHD; Gender
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Coitus | interventions — Nicotine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 4 (Experimental)
  Interventions: Drug: Nicotine; Other: Placebo

INTERVENTIONS:
Drug: Nicotine — 21 mg nicotine patches for smokers for 2 days
  7 mg nicotine patches for nonsmokers for 2 days
Other: Placebo — Placebo Patch

SUMMARY:
Attention deficit hyperactivity disorder (ADHD) is characterized by inattention, impulsivity, and hyperactivity that are frequently treated with stimulant medications such as Ritalin. Many people with ADHD smoke. The smoking prevalence rates are estimated to be 40% in adults with ADHD compared to 20% in the general population. People with ADHD have also more difficulty to quit smoking. Only 29% of smokers with ADHD quit smoking compared to 48.5% of smokers in the general population. Nicotine is a stimulant, which may have properties similar to stimulant medications (e.g., Ritalin) used to treat ADHD. Nicotine may increase attention and reduce hyperactivity and impulsivity and, thus, may regulate behavior in individuals with ADHD. Alleviating the symptoms of ADHD and increasing cardiovascular activity through smoking may mimic the effects of stimulant medications and can be a form of self-medication.

The major objective of the study was to examine the effects of nicotine on ADHD symptoms, moods, and cardiovascular activity. The study investigated the effects of nicotine patches on behavioral regulation in adult smokers and nonsmokers with ADHD. Smokers and nonsmokers with ADHD participated in two conditions: (1) nicotine patch and (2) placebo patch. During each condition, symptoms, moods, and side effects were assessed for 2 days during waking hours. An electronic handheld diary, programmed to prompt the participant twice per hour, recorded ADHD symptoms (e.g., difficulty concentrating, impulsivity, etc.), negative moods (e.g., anger, stress), and nicotine side effects (nausea, dizziness). Heart rate and blood pressure were recorded with lightweight ambulatory monitors to indicate cardiovascular activity. Results provided information about the effects of nicotine patches on behavioral regulation in adult smokers and nonsmokers with ADHD.

The inclusion of nonsmokers was important to clarify whether the effects of nicotine on smokers was due to smoking withdrawal. The findings help explain the increased smoking prevalence rates and reduced quit rates associated with ADHD. Knowledge about nicotine's effects on behavioral regulation can help to develop successful smoking cessation programs for individuals with ADHD. The findings on cardiovascular activity may help determine the potential risk for cardiovascular disease in smokers and nonsmokers with ADHD. The study contributed to understanding nicotine's effects on behavioral regulation in a highly vulnerable population such as people with ADHD.

ELIGIBILITY:
Inclusion Criteria:

* An age of 18 to 45 years
* A history of ADHD
* Current diagnosis of ADHD according to clinical criteria
* Being a smoker who smokes at least 10 cigarettes per day with 0.5 mg of nicotine per cigarette; OR
* Being a nonsmoker who has been abstaining from smoking and other nicotine products for the last 2 years

Exclusion Criteria:

* Treatment for any chronic illness such as heart disease, irregular heartbeat, high blood pressure, diabetes, skin allergies or skin diseases, including psoriasis or eczema, even if currently controlled by medication
* Current pregnancy, as measured by a pregnancy test (Clear Blue Easy, Unipath, Bedford, UK), or planning to become pregnant within the next 6 months. These individuals will not be included as the nicotine patch may cause harm to the unborn fetus
* Nursing mothers, or women who have breastfed within the last 12 months
* Non-English speaking people, because the majority of measurements used in the study have not been validated in languages other than English
* Current major depressive episode according to clinical criteria
* Concurrent psychiatric psychoactive medication within the past 12 months
* Active substance abuse within the past 12 months

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2005-08; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean G Gehricke, Ph.D., Principal Investigator — University of California, Irvine
Locations (1):
- Department of Pediatrics, Irvine, California, United States

REFERENCES:
- [Result] Gehricke JG, Hong N, Whalen CK, Steinhoff K, Wigal TL. Effects of transdermal nicotine on symptoms, moods, and cardiovascular activity in the everyday lives of smokers and nonsmokers with attention-deficit/hyperactivity disorder. Psychol Addict Behav. 2009 Dec;23(4):644-55. doi: 10.1037/a0017441. PMID 20025370

RESULTS

PARTICIPANT FLOW:
Groups:
- Smokers: In a modified within-group cross-over, smokers received 21 mg/day nicotine patches for two consecutive days and matching placebo patches for two consecutive days, with the order counterbalanced across participants.
- Nonsmokers: In a modified within-group cross-over, nonsmokers received 7 mg/day nicotine patches for two consecutive days and matching placebo patches for two consecutive days, with the order counterbalanced across participants.
Period: Overall Study
Arm/Group | Smokers | Nonsmokers
Started | 40 | 38
Nicotine Patches and Placebo Patches | 25 | 27
Completed | 25 | 27
Not Completed | 15 | 11
Not completed — scheduling conflicts | 15 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Smokers | Nonsmokers | Total
Number analyzed (Participants) | 40 | 38 | 78
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 40 | 38 | 78
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 25 (7) | 28 (8) | 27 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 13 | 22
  Male | 31 | 25 | 56
Region of Enrollment [Number; unit: participants]
  United States | 40 | 38 | 78

OUTCOME MEASURES:

1. Primary Outcome: ADHD Symptoms
Description: Mean percentage of endorsement for each electronic diary item (percent of 'yes' on an item) during 2 days on nicotine patches versus 2 days placebo patches
Time Frame: 4 days
Population: Per protocol, average ADHD symptoms, cardiovascular activity and moods during nicotine compared to placebo.
Measure: Mean (Standard Error); unit: Percent of item endorsement
Groups:
- Nicotine Patches: Smokers received 21 mg/day patches for two consecutive days and nonsmokers received 7 mg/day nicotine patches for two consecutive days.
- Placebo Patches: Smokers and nonsmokers received placebo patches for two consecutive days.
Arm/Group | Nicotine Patches | Placebo Patches
Number analyzed (Participants) | 52 | 52
Percent of item endorsement
  Difficulty concentrating | 71.2 (4.0) | 78.4 (3.4)
  Forgetfulness | 47.4 (4.0) | 55.5 (4.4)
  Restlessness | 71.8 (3.9) | 78.5 (3.2)
  Impatience | 72.3 (4.2) | 79.4 (3.7)
  Impulsivity | 61.8 (4.7) | 71.5 (3.9)
Statistical Analysis 1: Comparison: Nicotine Patches vs Placebo Patches; 2 (nicotine versus placebo) x 2 (smokers versus nonsmokers) ANOVA for each diary item; Test type: Superiority or Other; p < 0.025, ANOVA — Adjusted for multiple comparisons

2. Secondary Outcome: Blood Pressure
Description: Average blood pressure during 2 days on nicotine patches versus 2 days on placebo patches
Time Frame: 4 days
Measure: Mean (Standard Deviation); unit: mm HG
Arm/Group | Nicotine Patches | Placebo Patches
Number analyzed (Participants) | 52 | 52
mm HG
  Systolic Blood Pressure | 134 (17) | 131 (16)
  Diastolic Blood Pressure | 81 (11) | 78 (12)
Statistical Analysis 1: Comparison: Nicotine Patches vs Placebo Patches; 2 (nicotine versus placebo) x 2 (smoker versus nonsmoker) ANOVA; Test type: Superiority or Other; p < 0.025, ANOVA

3. Primary Outcome: Negative Moods
Description: as for outcome 1
Time Frame: 4 days
Measure: Mean (Standard Error); unit: Percent of item endorsement
Arm/Group | Nicotine Patches | Placebo Patches
Number analyzed (Participants) | 52 | 52
Percent of item endorsement
  Anger | 60.0 (4.5) | 71.4 (4.1)
  Nervousness | 69.7 (4.1) | 77.1 (3.4)
  Stress | 66.9 (4.4) | 74.2 (3.9)
Statistical Analysis 1: Comparison: Nicotine Patches vs Placebo Patches; 2 (nicotine versus placebo) x 2 (smokers versus nonsmokers) ANOVA for each diary item; Test type: Superiority or Other; p < 0.025, ANOVA — Adjusted for multiple comparisons

4. Primary Outcome: Side Effects
Description: as for outcome 1
Time Frame: 4 days
Measure: Mean (Standard Error); unit: Percent of item endorsement
Arm/Group | Nicotine Patches | Placebo Patches
Number analyzed (Participants) | 52 | 52
Percent of item endorsement
  Nausea | 37.7 (3.5) | 30.7 (3.6)
  Dizziness | 33.5 (3.2) | 33.8 (3.5)
Statistical Analysis 1: Comparison: Nicotine Patches vs Placebo Patches; 2 (nicotine versus placebo) x 2 (smokers versus nonsmokers) ANOVA for each diary item; Test type: Superiority or Other; p < 0.025, ANOVA — Adjusted for multiple comparisons

ADVERSE EVENTS:
Arm/Group | Smokers | Nonsmokers
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/27
Other Adverse Events (participants affected / at risk) | 0/25 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No